CLINICAL TRIAL: NCT07348146
Title: Hand-Sewn vs. Stapled Anastomosis in SADI-S: A Prospective Randomized Trial of Early Postoperative Complications.
Brief Title: Hand-Sewn vs. Stapled Anastomosis in SADI-S: Early Postoperative Complications.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Abdelsalam M, Associate Professor of General and Laparoscopic Surgery, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Stapled SADIs 082025
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Metabolic Surgery; Obesity & Overweight
Keywords: Stapled versus Hand-sewn Technique; SADI-s; Metabolic Bariatric Surgery
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hand-sewn Single Anastomosis Duodeno-Ileal Sleeve (SADI-S) (Active Comparator)
  Interventions: Procedure: Hand-sewn Single Anastomosis Duodeno-Ileal Sleeve (SADI-S)
- Stapled Single Anastomosis Duodeno-Ileal Sleeve (SADI-S) (Active Comparator)
  Interventions: Procedure: Stapled Single Anastomosis Duodena-ileal Sleeve

INTERVENTIONS:
Procedure: Hand-sewn Single Anastomosis Duodeno-Ileal Sleeve (SADI-S) — Arm 1 - Hand-sewn Duodeno-Ileal Anastomosis Following sleeve gastrectomy, a hand-sewn duodeno-ileal anastomosis is performed in two layers, with the inner layer constructed using absorbable barbed sutures and the outer reinforcing layer using absorbable monofilament sutures. Approximately 300 cm of the distal ileum from the ileocecal junction is used for the anastomosis. All procedures are performed by the same surgeon following a standardized operative protocol.
  Arms: Hand-sewn Single Anastomosis Duodeno-Ileal Sleeve (SADI-S)
Procedure: Stapled Single Anastomosis Duodena-ileal Sleeve — Arm 2 - Stapled Single Anastomosis Duodena-ileal Sleeve Following sleeve gastrectomy, a stapled duodeno-ileal anastomosis is created using endoscopic linear stapling devices, followed by closure of the enterotomy in a single layer using absorbable barbed sutures. Approximately 300 cm of the distal ileum from the ileocecal junction is used for the anastomosis. All procedures are performed by the same surgeon following a standardized operative protocol.
  Arms: Stapled Single Anastomosis Duodeno-Ileal Sleeve (SADI-S)

SUMMARY:
This study aims to compare the stapled and handsewn techniques of duodeno-ileal anastomosis in SADI-S regarding short-term outcomes in the form of anastomotic leak rate and anastomotic stricture rate, operative time, post-operative hospital stay, and complication rate (Clavien-Dindo≥ II).

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-70
2. Patients who will undergo SADI-S surgery

Exclusion Criteria:

1. Patients with severe medical conditions such as heart failure and interstitial lung disease.
2. Patients with short bowel
3. Patients with severe GERD
4. Patients with cognitive and intellectual impairment with poor compliance to treatment and dietary supplements
5. Difficulty in intraoperative bowel measurement, i.e., extensive adhesions.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Intestinal Injury | One month after surgery
Anastomotic Leak Rate | one month after the surgery
Post operative Bleeding | One month after surgery
Anastomotic Stircture | Six months after surgery
Operative Time | Immediately after surgery

SECONDARY OUTCOMES:
Weight loss | Six months after surgery
Length of Hosptial Stay | One month after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy Medical School, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kshirsagar VV, Mp H. A Comparative Study of Hand-Sewn and Stapled Anastomosis in Gastrointestinal Surgeries. Cureus. 2024 Oct 11;16(10):e71264. doi: 10.7759/cureus.71264. eCollection 2024 Oct. PMID 39525136
- [Background] Ebinuma S, Kunisawa S, Fushimi K, Ichikawa N, Yoshida T, Homma S, Taketomi A, Imanaka Y. Comparative retrospective study on surgical outcomes of hand-sewn anastomosis versus stapling anastomosis for colectomy using a nationwide inpatient database in Japan with propensity score matching. Ann Gastroenterol Surg. 2024 Oct 11;9(2):379-388. doi: 10.1002/ags3.12870. eCollection 2025 Mar. PMID 40046528
- [Background] Pennestri F, Sessa L, Prioli F, Salvi G, Gallucci P, Ciccoritti L, Greco F, De Crea C, Raffaelli M. Single anastomosis duodenal-ileal bypass with sleeve gastrectomy (SADI-S): experience from a high-bariatric volume center. Langenbecks Arch Surg. 2022 Aug;407(5):1851-1862. doi: 10.1007/s00423-022-02501-z. Epub 2022 Mar 29. PMID 35352174
- [Background] O'Brien PE, Hindle A, Brennan L, Skinner S, Burton P, Smith A, Crosthwaite G, Brown W. Long-Term Outcomes After Bariatric Surgery: a Systematic Review and Meta-analysis of Weight Loss at 10 or More Years for All Bariatric Procedures and a Single-Centre Review of 20-Year Outcomes After Adjustable Gastric Banding. Obes Surg. 2019 Jan;29(1):3-14. doi: 10.1007/s11695-018-3525-0. PMID 30293134
- [Background] Lazzati A, Bechet S, Jouma S, Paolino L, Jung C. Revision surgery after sleeve gastrectomy: a nationwide study with 10 years of follow-up. Surg Obes Relat Dis. 2020 Oct;16(10):1497-1504. doi: 10.1016/j.soard.2020.05.021. Epub 2020 May 29. PMID 32636173
- [Background] Aleassa EM, Hassan M, Hayes K, Brethauer SA, Schauer PR, Aminian A. Effect of revisional bariatric surgery on type 2 diabetes mellitus. Surg Endosc. 2019 Aug;33(8):2642-2648. doi: 10.1007/s00464-018-6541-1. Epub 2018 Oct 19. PMID 30341657